CLINICAL TRIAL: NCT03920709
Title: Analysis of the Nasal Mucosal Immune Response in HIV Infection
Acronym: HYSOPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pasteur Institute of Paris (Unknown)
Responsible Party: Sponsor
Other Study IDs: HYSOPE
Record Dates: First submitted 2019-01-10; First posted 2019-04-19 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample and nasal mucosa
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic HIV-1 infected subjects : 50 Viremic subjects: plasma HIV RNA > 500 copies/mL, treatment-naive or treated (failing) regardless of the cause of persistent viremia
  Interventions: Other: Blood sample and Nasal swabs (right an left) samples
- Chronic HIV-1 infected subjects : 50 Treated Aviremic subjects: < 50 copies/mL under treatment for at least 12 months
  Interventions: Other: Blood sample and Nasal swabs (right an left) samples
- Chronic HIV-1 infected subjects :10 Spontaneous Controllers: from the ANRS CO21 CODEX Cohort or not (5 last viral loads < 400 copies /ml)
  Interventions: Other: Blood sample and Nasal swabs (right an left) samples

INTERVENTIONS:
Other: Blood sample and Nasal swabs (right an left) samples — Nasal swabs (right and left) will be performed (FLOQSwabTM)
  Blood samples of 20 mL EDTA will be taken in addition to the current care report

SUMMARY:
The principal objective is to define and compare the viral reservoir, mucosal immune responses and the microbiota of different HIV infection stages; viremic, aviremic (under treatment), natural elite controllers; The secondary objective is to compare the mucosal immune response and microbiota of HIV patients with the healthy control population of Milieu Interieur;

DETAILED DESCRIPTION:
Although antiretroviral therapy (ART) efficiently suppresses viral replication HIV persists in CD4+ T cells in a form that is neither targeted by the immune system nor by ART, the complete eradication of replication competent HIV or the establishment of a long term remission state in infected individuals represents an outstanding challenge.

The persistence of reservoirs has been mainly linked to the survival and clonal expansion of pools of long lived infected memory CD4+ T cells and to low level viral replication in tissues where ART penetration may be incomplete. One such tissue may be mucosal surfaces which are challenging to study in human populations.

As part of the Milieu Interieur project, coordinated by Institut Pasteur, investigators have developed and validated a standardized approach for sampling the nasal mucosa. From this simple sampling procedure it is possible to analyze both the local mucosal host immune response at the proteomic and metabolomic level, and also the mucosal microbial flora.

As part of Milieu Interieur investigators have defined these diverse phenotypes for a subset of donors and are currently extending the analysis to the 1,000 healthy donors cohort that will give reference range values for the nasal mucosa.

Investigators wish to compare with relevant patient groups, in particular HIV infected individuals to see how infection, treatment, and natural host control may differentially impact the mucosal immune response and viral reservoir

ELIGIBILITY:
Inclusion Criteria:

* Chronic HIV-1 infected subjects followed in Department of Internal Medicine and Clinical Immunology in Bicetre Hospital
* Healthy male or female aged between 20 and 69 (included) years
* Whatever the clinical status and the lymphocytes T CD4+
* Patients treatment-naive or under ARV treatment whatever the molecules
* 3 groups of patients, according to their HIV1 viral loads

  * Virémic : viral load > 500 copies/mL, treatment-naive or treated (failing) regardless of the cause of persistent viremic
  * No Viremic : < 50 copies/ml under treatment at least from 12 months
  * Spontaneous Controllers from the Codex Cohort (Controllers cohort from ANRS) or not with the following inclusion criteria Chronic HIV-1 infected subjects since 5 years, asymptomatic With 5 last viral loads < 400 copies /mL Whatever the lymphocytes T CD4 rates Naive of treatment except transient treatment for prevention of mother-to-child transmission
* Subject considered to be free on the day of study of an acute condition or infection that may interfere with the results of the study, based on the clinical examination performed by the investigator
* Caucasian and Sub Saharan patients -18,5 ≤ BMI ≤ 32 kg/m²
* Subjects who, according to the investigator, can and will comply with the requirements of the protocol and are available for the scheduled visit at the investigational site. Ability to give their informed consent in writing
* Affiliated to the French social security or assimilated regimens

Exclusion Criteria:

Participation in another clinical study in the last 3 months

* Travel in (sub-) tropical countries within the last 3 months
* Pregnant women
* Infectious diseases:

  * Acute opportunistic or not, current or past infection, within the last 3 months as determined by the PI
  * Ear temperature ≥ 38.4 ° C on the day of inclusion
  * Subject currently receiving or having received in the last 3 months antibiotics or nasal, intestinal or respiratory antiseptics
* Severe/chronic/recurrent pathological conditions, among them:

  * Past or present diagnosed cancer, lymphoma, leukemia to the exception of: Persons with a history of cancer who are disease-free without treatment for 5 years or more
  * Women who are disease free for 3 years or more after treatment for breast cancer and receiving long-term prophylactic tamoxifen
  * Cutaneous or cervical basal cell carcinoma
  * Personal history of organ transplant
  * Congenital or acquired immune deficiency (any confirmed or suspected immunosuppressive or immunodeficient condition, including history of HIV infection)
  * Personal history of auto-immune diseases requiring or having previously required treatment (e.g. Rheumatoid Arthritis, Systemic Lupus Erythematosus, Sarcoidosis, Ankylosing Spondylitis, Autoimmune Hemolytic Anemia, Autoimmune Thrombocytopenic Purpura, Crohn's Disease, Psoriasis, Scleroderma, Wegener's Granulomatosis,Type I Diabetes, Thyroiditis,….)
  * Splenectomy
  * Acute or chronic, clinically significant, as determined by the investigator, pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory
  * Chronic renal impairment as defined by Renal Insufficiency: GFR<60 mL/min/1.73 m² (National Kidney Foundation (2002)
  * History of clinically significant, as determined by the investigator, neurological disorder or seizures
  * Any physical activity within 8 hours before the visit
  * Any significant disorder of coagulation or treatment with warfarin derivatives (AVK or ACO)or heparin or antiplatelet medications within 2 months preceding inclusion
* Severe acute/chronic allergy

  * Severe Asthma defined as asthma requiring a combination of two or more controller therapies (e.g. medium or high dose inhaled glucocorticosteroid and long-acting inhaled beta-2 agonist) or requiring oral glucocorticosteroids (GINA),
  * Severe insect bite allergy with history of giant urticaria, Quincke edema or anaphylactic shock
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within the 6 months prior to the inclusion. For corticosteroids, this will mean a dose equivalent to 20 mg/day of prednisone or equivalent for > 2 weeks (inhaled and topical steroids allowed)
* Chronic administration of NSAIDs, including aspirin: prolonged intake (> 2 weeks) within 6 months before study
* Receipt of blood products or immunoglobulins within 3 months prior the inclusion or planning to receive blood products or immunoglobulins during the study
* Hemoglobin measurement less than 10.0 g/dL for women and less than 11.5 g/dL for men
* Platelet count less than 120.000/mm3
* ALAT and/or ASAT > 3 times the upper limit of the norm (ULN)
* Receipt of any vaccination 3 months before the inclusion
* Alcohol abuse (more than 50 g of pure ethanol per day: for example, more than 4 x 150 mL glasses of wine, more than 4 x 250 mL glasses of beer, more than 4 x 40 mL glasses of high alcohol content drinks
* Illicit drug use or substance abuse within 3 months prior to inclusion

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 110 patients followed in Department of Internal Medicine and Clinical Immunology Bicetre Hospital APHP Chronic HIV-1 infected subjects
  * 50 Viremic subjects : plasma HIV RNA > 500 copies/mL, treatment-naive or treated (failing) regardless of the cause of persistent viremia
  * 50 Treated Aviremic subjects : < 50 copies/mL under treatment for at least 12 months
  * 10 Spontaneous Controllers from the ANRS CO21 CODEX Cohort or not (5 last viral loads < 400 copies /ml)
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of HIV p24 levels in the supernatants of nasal mucosa | through study completion, an average of 2 years
  Measurement of HIV p24 levels in the supernatants of nasal mucosa in HIV-infected patients in the 3 groups

SECONDARY OUTCOMES:
HIV p24 levels in the supernatants and in the pellets of the nasal mucosa in HIV-infected patients | through study completion, an average of 2 years
  Quantification of HIV p24 levels in the supernatants and in the pellets of the nasal mucosa
Assessement of the microbiome in the nasal mucosa | through study completion, an average of 2 years
  Description of nasal mucosa microbiome diversity in the nasal mucosa of HIV-infected patients, and comparison with control subjects from the Milieu intérieur Cohort

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Goujard, Pr, Principal Investigator — AP-HP Hôpital Bicêtre
Locations (1):
- Pr GOUJARD Cécile, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be entered electronically via a web browser in Electronic Case Report Form Data will be analysed by Pasteur Institute of Paris with the biological results
Supporting Information: CSR, Analytic Code
Time Frame: At the end of the study
Access Criteria: The persons responsible for the quality control of clinical studies (the French Public Health Code) will take all necessary precautions to ensure the confidentiality of information relating to the research, the participants and in particular their identity and the results obtained. These persons, as well as the investigators themselves, are bound by professional secrecy. During and after the research, all data collected about the participants and sent to the Pasteur Institute of Paris by the investigators will be anonymized. Under no circumstances will the names and addresses of the participants be shown. The sponsor will ensure that each participant has agreed in writing for any personal information about him or her which is strictly necessary for the quality control of the study to be accessed Identification of the person responsible and the location for data processing. Statistical analysis will be performed by scientist and IPP bio-informatician within the research units involved.